CLINICAL TRIAL: NCT05431127
Title: High-dose Inspiratory Muscle Training (IMT) in Late-onset Pompe Disease (LOPD)
Brief Title: High Dose Inspiratory Muscle Training in LOPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00109392
Record Dates: First submitted 2022-06-21; First posted 2022-06-24 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-05

CONDITIONS: Late-Onset Pompe Disease; Lysosomal Disease
Keywords: LOPD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High Dose Inspiratory Muscle Training (Other): Inspiratory Muscle Training 3 times a week over 26 weeks
  Interventions: Device: IMT therapy using the Pr02 mobile device

INTERVENTIONS:
Device: IMT therapy using the Pr02 mobile device — Inspiratory Muscle Training using a device used to measure and increase respiratory strength and performance through resisted breathing exercises.

SUMMARY:
Study Objectives: 1) assess the safety and feasibility of high-dose inspiratory muscle training (IMT) delivered remotely in Late-onset Pompe Disease (LOPD) and 2) determine its effects on respiratory and patient-reported outcomes.

DETAILED DESCRIPTION:
This study aims to develop treatments that enhance respiratory strength and function to provide meaningful clinical improvements for people with LOPD. Identification of a cost-effective adjunctive intervention to address respiratory weakness remains critical to reduce disease burden, ease activity limitations and participation restrictions, and improve health-related quality of life. The proposed study will provide a high-dose inspiratory muscle training (IMT) stimulus to enhance treatment efficacy and efficiency. Our hypothesis is that high-dose IMT is necessary to produce meaningful changes in respiratory muscle strength and other outcomes in participants with LOPD.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Confirmed diagnosis of LOPD
* MIP >50% of predicted for sex and age
* Stable on current Pompe disease treatment regimen >6 months
* Able to follow directions for study participation
* Access to computer and smartphone/tablet with reliable internet connection for video visits and sensor-based respiratory technologies

Exclusion Criteria:

* Presence of medical comorbidities that prevent meaningful study participation (e.g., COPD GOLD III-IV, significant mental illness, dementia)
* Use of continuous invasive or non-invasive ventilation while awake
* Prior history of gene therapy for LOPD
* Inability to give legally effective consent
* Inability to read and understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Change in maximum inspiratory pressure (MIP) | Baseline, week 15, week 30
  Change pre-test to post test, measured in cm H20

SECONDARY OUTCOMES:
Change in maximum expiratory pressure (MEP) | Baseline, week 15, week 30
  Change pre-test to post test, measured in cm H20
Change in inspiratory power curve (IPC) | Baseline, week 15, week 30
  Change pre-test to post test, measured in pressure-time units (PTUs)
Change in inspiratory duration (ID) | Baseline, week 15, week 30
  Change pre-test to post test, measured by duration in seconds
Change in fatigue index test score (FIT) | Baseline, week 15, week 30
  Change pre-test to post test, a proprietary measure which quantifies propensity to inspiratory muscle fatigue based upon the relationship between inspiratory capacity and demand using the following equation: (IPC [in Watts] x MID) / (Power500 x T500), where Power500 = power expended to inspire a mass of 500 mL air and T500 = time when mass of inspired air=500 mL at sea level
Change in forced vital capacity (FVC) | Baseline, week 15, week 30
  Change pre-test to post-test, measured in liters using a portable hand-held spirometer
Change in forced expiratory volume over 1 second (FEV1) | Baseline, week 15, week 30
  change pre-test to post-test, measured in liters per second using a portable hand-held spirometer
Change in peak expiratory flow (PEF) | Baseline, week 15, week 30
  change pre-test to post-test, measured in liters per second using portable hand-held spirometer
Change in inspiratory phase duration (IPD) | Baseline, week 15, week 30
  change pre-test to post-test, measured in seconds
Change in inspiratory peak flow (IPF) | Baseline, week 15, week 30
  Change pre-test to post-test, measured in liters per second
Change in compression phase duration (CPD) | Baseline, week 15, week 30
  Change pre-test to post-test, measured in seconds
Change in expiratory phase rise time (EPRT) | Baseline, week 15, week 30
  Change pre-test to post-test, measured in liters per second
Change in cough volume acceleration (CVA) | Baseline, week 15, week 30
  Change pre-test to post-test, measured by EPF/EPRT
Change in fatigue | Baseline, week 15, week 30
  Change pre-test to post-test, measured by Fatigue Severity Scale (FSS) survey completion, using a 7 point ordinal scale where a rating of 1 indicates strong disagreement and a rating of 7 indicates strong agreement.
Change in impact of fatigue on quality of life (QOL) | Baseline, week 15, week 30
  Change pre-test to post-test, measured by Modified Fatigue Impact Scale (MFIS) survey completion using a score of 0 (never affected) to 4 (almost always affected). The total score ranges from 0 to a maximum of 84. Higher scores indicate greater impact of fatigue on quality of life.
Change in daytime sleepiness | Baseline, week 15, week 30
  Change pre-test to post-test, measured by Epworth Sleepiness Scale (ESS) survey completion using a 0 to 3 ordinal scale in which 0=no chance of dozing, 1=slight chance of dozing, 2= moderate chance of dozing, and 3=high chance of dozing. Scores are summed to obtain total ESS score where a score >10 reflects excessive daytime sleepiness.
Change in sleep quality | Baseline, week 15, week 30
  Change pre-test to post-test, measured by Pittsburgh Sleep Quality Index (PSQI) survey completion. The PSQI is a 9-question, 19-item instrument. Items 1 to 4 are open-ended questions (customary bedtime, length of time to fall asleep). Items 5 to 8 (including the 10 questions comprising item 5) are sleep symptoms which are rated as to their frequency using an ordinal scale: 0=not occurring in the last month, 1=less than once a week, 2=once or twice a week, and 3=three or more times a week. Item 9 is a rating of overall sleep quality over the past month using a 0 to 3 ordinal scale: 0=very good; 1=fairly good; 2= fairly bad; and 3=very bad. Scores from the 19-items are combined according to standard scoring criteria to obtain a Global PSQI score. Scores >5 indicate reduced sleep quality.
Change in respiratory symptoms | Baseline, week 15, week 30
  Change pre-test to post-test, measured by Respiratory Symptoms Questionnaire (RSQ) completion using a 0-3 scale where a higher score indicates worse symptoms.
Change in motor performance | Baseline, week 15, week 30
  Change pre-test to post-test, measured by Rotterdam Handicap Scale (RHS) survey completion using a ranging scale of 1 - 4 where 1 = unable to fulfil the task or activity and 4 = complete fulfillment of the task or activity. Scores are summed and range from 9-36.
Change in health-related quality of life | Baseline, week 15, week 30
  Change pre-test to post-test, measured by Short Form 36 (SF-36) survey completion where physical and mental component summary scales (PCS and MCS) are calculated from the subscales and transformed to a normalized T-score with a mean of 50 and a standard deviation of 10. Higher scores represent better health-related quality of life.
Change in ability to communicate | Baseline, week 15, week 30
  Change pre-test to post-test, measured by Communicative Participation Item Bank-Short From (CPIB-10) survey completion using a 4-point scale (not at all=3, a little=2, quite a bit=1, very much=0). Item scores are added to obtain the summary score which ranges from 0-30. This can be transformed into a standard T score (mean=50, SD=10). Higher scores represent less interference in communication participation.
Change in voice quality | Baseline, week 15, week 30
  Change pre-test to post-test, measured by Voice Handicap Index (VHI-10) survey completion using a 5-point scale (0=never, 1=almost never, 2=sometimes, 3=almost always, 4=always). Item responses are added to obtain a total score (values >11 abnormal) with higher scores indicating greater perception of voice-related handicap.
Change in swallowing symptoms | Baseline, week 15, week 30
  Change pre-test to post-test, measured by Eating Assessment Tool (EAT-10) survey completion using a 5-point scale (0=no problem, 4=severe problem). Item responses are added to obtain a total score (values >3 abnormal) with higher scores indicating greater severity of swallowing symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Harrison Jones, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No